CLINICAL TRIAL: NCT03342807
Title: Randomized, Controlled, Multicenter Studies of the Effects of Intravenous Administration of Insulin and Plasma Exchange on Triglyceride Levels in Early Stage of Hypertriglyceridemia-induced Pancreatitis
Brief Title: Intravenous Administration of Insulin and Plasma Exchange on Triglyceride Levels in Early Stage of Hypertriglyceridemia-induced Pancreatitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: First Hospitals affiliated to the China PLA General Hospital (Other Government); Nanjing General Hospital (Unknown); Fujian Provincial Hospital Emergency Center (Unknown); First Affiliated Hospital, Sun Yat-Sen University (Other); Jinhua Central Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); First Affiliated Hospital of Kunming Medical University (Other); Tianjin Medical University General Hospital (Other); The First Hospital of Hebei Medical College (Unknown); The First Affiliated Hospital with Nanjing Medical University (Other); Shenzhen Baoan District People 's Hospital (Unknown); The General Hospital of Shenyang Military (Unknown); Cangzhou Center Hospital (Unknown); Wuxi Third People 's Hospital (Unknown); General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HTG-AP-Insulin
Record Dates: First submitted 2017-11-05; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-08

CONDITIONS: Pancreatitis, Acute; Hypertriglyceridemia
Keywords: Hypertriglyceridemia-induced acute pancreatitis; insulin; triglyceride; treatment
MeSH Terms: conditions — Pancreatitis; Hypertriglyceridemia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group Insulin (Experimental)
  Interventions: Drug: Insulin
- Group Aphesis (Experimental)
  Interventions: Device: Aphesis

INTERVENTIONS:
Drug: Insulin — Insulin infusion for subjects in Group Insulin.
  Arms: Group Insulin
Device: Aphesis — Aphesis for subjects in Group Aphesis.
  Arms: Group Aphesis

SUMMARY:
To investigate an economical and effective way to reduce the level of serum triglyceride in patients with hypertriglyceridemia-induced acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 to 80 years old;
2. abdominal pain consistent with AP;
3. serum amylase and / or lipase activity is at least 3 times higher than the normal upper limit;
4. abdominal imaging consistent with AP imaging changes.
5. severe hyperlipidemia "fasting serum TG> 1,000 mg/dL (11.2mmol/L)";
6. except for other AP causes, such as cholelithiasis, alcohol, drugs and so on.

Exclusion Criteria:

1. other etiologies other than hyperlipidemia leading to AP;
2. fasting serum TG less than 1,000 mg / dL (11.2mmol / L);
3. acute lipid-induced pancreatitis at the same time combined with other etiologies of acute pancreatitis.
4. the existence of plasma replacement contraindications: serious allergies to plasma, human serum albumin, heparin and others; the existence of mental disorders; unstable heart or cerebral infarction; intracranial hemorrhage or severe cerebral edema associated with hernia.
5. without informed consent, the patient refused to plasma replacement, and other circumstances may bring significant bias.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-11 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
serum TG | every 4 hours in first 3 days
  Elimination of serum triglyceride.

REFERENCES:
- [Derived] Song X, Shi D, Cui Q, Yu S, Yang J, Song P, Walline J, Xu J, Zhu H, Yu X. Intensive insulin therapy versus plasmapheresis in the management of hypertriglyceridemia-induced acute pancreatitis (Bi-TPAI trial): study protocol for a randomized controlled trial. Trials. 2019 Jun 18;20(1):365. doi: 10.1186/s13063-019-3498-x. PMID 31215460